CLINICAL TRIAL: NCT05711745
Title: Effects of Myofascial Induction Therapy on Ankle Pressure Pain and Ankle Range of Motion in Latent Trigger Points of the Gastrocnemius Muscle. A Clinical Trial.
Brief Title: Effects of Myofascial Induction Therapy on Pressure Pain and Ankle Range of Motion.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayuben Private Clinic (Other)
Responsible Party: Principal Investigator, EVA MARIA MARTÍNEZ JIMENEZ, Fisioterapist responsible area, Mayuben Private Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2911202021420A
Record Dates: First submitted 2023-01-16; First posted 2023-02-03 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Fascia; Trigger Point Pain, Myofascial; Range of Motion; Pain
MeSH Terms: conditions — Myofascial Pain Syndromes; Pain

STUDY DESIGN:
Intervention Model Description: A pre-post study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Myofascial induction in gastrocnemius (Experimental): A 3-pass superficial leg glide technique was applied first and then 5 minutes of the deep calf myofascial induction technique as described by Pilat.
  Interventions: Procedure: Calf myofascial technique

INTERVENTIONS:
Procedure: Calf myofascial technique — A 3-pass superficial leg glide technique was applied first and then 5 minutes of the deep calf myofascial induction technique as described by Pilat.

SUMMARY:
In this study, it will be assessed if there are changes in ankle dorsiflexion and pressure pain after performing the myofascial induction technique in the calf.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with no pain and with 18 to 30 years old.

Exclusion Criteria:

* (1) Diagnosis of lower limb injury, including any tendinopathy, bursitis, ligamentous involvement or fasciitis ,
* (2) history of lower limb surgery ,
* (3) participants were required not to have undergone ankle stretching or any other treatment,
* (4) diabetes due to possible alteration of arterial distal circulation,
* (5) deformities of the toes, such as hammer toes and hallux valgus. All subjects signed an informed consent form before participating in the study

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2023-02-08 (Actual); Study Completion 2023-02-09 (Actual)

PRIMARY OUTCOMES:
Pressure pain threshold | Immediately before intervention.
  The pressure at which the patient begins to feel pain with pressure is measured 3 times with an algometer.It is measured in newtons
Range of motion with knee extended | Immediately before the intervention.
  The joint range is measured in dorsiflexion of the ankle joint with the knee extended under load and is measured with an inclinometer in degrees.Measured in grades.
Range of motion with knee flexed | Immediately before the intervention.
  The joint range is measured in dorsiflexion of the ankle joint with the knee flexed under load and is measured with an inclinometer in degrees. Measured in grades.
Pressure pain threshold | Immediately after the intervention.
  The pressure at which the patient begins to feel pain with pressure is measured 3 times with an algometer.It is measured in newtons
Range of motion with knee extended | Immediately after the intervention.
  The joint range is measured in dorsiflexion of the ankle joint with the knee extended under load and is measured with an inclinometer in degrees.Measured in grades.
Range of motion with knee flexed | Immediately after the intervention.
  The joint range is measured in dorsiflexion of the ankle joint with the knee flexed under load and is measured with an inclinometer in degrees.Measured in grades.

CONTACTS AND LOCATIONS:
Locations (1):
- Eva María Martinez Jiménez, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No